CLINICAL TRIAL: NCT05075746
Title: Retrospective Chart Review of enVista Toric 0.9D Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: BHC-RCR-001
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-09

CONDITIONS: Corneal Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- enVista Toric 0.9D intra ocular lens
  Interventions: Device: enVista Toric
- enVista non-Toric (spherical) intra ocular lens
  Interventions: Device: enVista non-Toric (spherical)

INTERVENTIONS:
Device: enVista Toric — enVista Toric IOL
  Groups: enVista Toric 0.9D intra ocular lens
Device: enVista non-Toric (spherical) — enVista non-Toric (spherical) IOL
  Groups: enVista non-Toric (spherical) intra ocular lens

SUMMARY:
The primary objective of this study is to evaluate the performance of the enVista Toric 0.9D vs non-Toric IOL.

DETAILED DESCRIPTION:
The performance of the enVista Toric IOLs will be compared with that of enVista non-Toric (spherical) IOL. At least 384 eyes (n= 192 per lens type) from 3-4 Canadian centers will be investigated.

This is a retrospective chart review for preoperative and postoperative data conducted at least 4 weeks after IOL implantation.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females subjects age 18 or older on the date of surgery
* Implant of enVista Toric IOL and/or enVista non-Toric (spherical) IOL in at least one eye
* Data available at least 4 weeks after IOL implantation
* Eyes must qualify for the 0.9D toric lens based on the Barrett Toric Calculator (flipped axis must be less than 0.2D) (https://ascrs.org/tools/barrett-toric-calculator)

  * Study eyes were implanted with the 0.9D toric lens
  * Control eyes were not implanted with the 0.9D toric lens and implanted with a spherical (non-toric) equivalent instead

Exclusion Criteria:

* History of uncontrolled or clinically significant ocular comorbidities for the treated eye(s) before the surgery (e.g., dry eyes, retinal pathology, etc.)
* BCDVA of 20/25 or worse for the treated eye(s) after the surgery
* Excessive IOL rotation > 10 degrees (Toric IOLs only) for the treated eye(s) after the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The performance of the enVista Toric IOLs will be compared with that of enVista non-Toric (spherical) IOL in patients with pre-op corneal astigmatism <1.0D. At least 384 eyes (n= 192 per lens type) from 3-4 Canadian centers will be investigated.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health
Locations (3):
- Canada (3):
  - Bausch Site 01, Calgary, Alberta
  - Bausch Site 03, Langley, British Columbia
  - Bausch Site 02, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | enVista Toric 0.9D Intra Ocular Lens | enVista Non-Toric (Spherical) Intra Ocular Lens
Started | 157; 192 Eyes | 145; 191 Eyes
Completed | 157; 192 Eyes | 145; 191 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | enVista Toric 0.9D Intra Ocular Lens | enVista Non-Toric (Spherical) Intra Ocular Lens | Total
Number analyzed (Participants) | 157 | 145 | 302
Number analyzed (Eyes) | 192 | 191 | 383
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (8.73) | 72.5 (8.44) | 71.6 (8.63)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 112 | 96 | 208
  Male | 80 | 95 | 175
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 25 | 49
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 99 | 96 | 195
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 64 | 66 | 130
Region of Enrollment [Number; unit: Eyes]
  Canada | 192 | 191 | 383

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction in Cylindrical Power of the Eye
Description: Reduction in the cylindrical power of the eye is defined as the difference between the magnitudes of the preoperative keratometric cylinder and the residual refractive cylinder (referenced to the corneal plane).
Time Frame: 4 weeks after IOL implantation
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Arm/Group | enVista Toric 0.9D Intra Ocular Lens | enVista Non-Toric (Spherical) Intra Ocular Lens
Number analyzed (Participants) | 157 | 145
Number analyzed (Eyes) | 192 | 191
Diopters | 0.432 (0.4468) | 0.071 (0.4073)

ADVERSE EVENTS:
Time Frame: 4 weeks after IOL implantation
Arm/Group | enVista Toric 0.9D Intra Ocular Lens | enVista Non-Toric (Spherical) Intra Ocular Lens
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/145
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/145
Other Adverse Events (participants affected / at risk) | 26/157 | 9/145
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | enVista Toric 0.9D Intra Ocular Lens (N=157) | enVista Non-Toric (Spherical) Intra Ocular Lens (N=145)
Posterior Capsule Opafication (Eye disorders) | 26 (31) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT05075746/Prot_SAP_000.pdf